CLINICAL TRIAL: NCT05127369
Title: Safety and Efficacy of Dental Pulp Mesenchymal Cells in the Treatment of Depression:
Brief Title: Clinical Study on the Safety and Efficacy of Dental Pulp Mesenchymal Cells in the Treatment of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CAR-T (Shanghai) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KT013HAN001
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Dental pulp mesenchymal cell injection (dose: 0.1u/kg) + fluoxetine hydrochloride
  Interventions: Drug: Dental pulp mesenchymal cell injection; Drug: fluoxetine hydrochloride capsule
- control group (Active Comparator): Dental pulp mesenchymal cell injection vehicle + fluoxetine hydrochloride capsule
  Interventions: Drug: Dental pulp mesenchymal cell vehicle; Drug: fluoxetine hydrochloride capsule

INTERVENTIONS:
Drug: Dental pulp mesenchymal cell injection — Dental pulp mesenchymal cell injection was administered intravenously on D1, D15 (2 weeks), D29 (4 weeks) and d43 (6 weeks); Fluoxetine hydrochloride capsule / simulant was administered orally daily.
  Arms: Test group
Drug: Dental pulp mesenchymal cell vehicle — Dental pulp mesenchymal cell vehicle was administered intravenously on D1, D15 (2 weeks), D29 (4 weeks) and d43 (6 weeks); Fluoxetine hydrochloride capsule / simulant was administered orally daily.
  Arms: control group
Drug: fluoxetine hydrochloride capsule — fluoxetine hydrochloride capsule

SUMMARY:
This is a single center phase I / II clinical trial. Randomized, blind and positive drug parallel control were used to evaluate the safety and effectiveness of dental pulp mesenchymal cell injection in the treatment of depression 8 weeks after administration

DETAILED DESCRIPTION:
This is a single center phase I / II clinical trial. Randomized, blind and positive drug parallel control were used to evaluate the safety and effectiveness of dental pulp mesenchymal cell injection in the treatment of depression 8 weeks after administration. The positive control drug was fluoxetine hydrochloride capsule with a dose of 40mg / day.The study included screening period (no more than 4 weeks), treatment period (8 weeks), and follow-up period (12 months).Subjects who met the inclusion criteria and did not meet the exclusion criteria were randomly assigned to the experimental group and the control group in the ratio of 1:1.During 8 weeks of treatment, subjects in the experimental group were given dental pulp mesenchymal cell injection + fluoxetine hydrochloride capsule simulant; The subjects in the control group were given dental pulp mesenchymal cell injection vehicle + fluoxetine hydrochloride capsule. During the treatment period, dental pulp mesenchymal cell injection / vehicle was injected intravenously for 4 times at an interval of 2 weeks (once at 0, 2, 4 and 6 weeks respectively); At the same time, fluoxetine hydrochloride capsule / simulant was taken orally every day during the treatment period.The efficacy and safety were evaluated 2 weeks after intravenous administration (visit and evaluation at 2, 4, 6 and 8 weeks respectively). Safety telephone follow-up was conducted 4 weeks (10th week), 6 months and 12 months after the last intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form, the age of 18 ≤ 60, regardless of gender.
2. 18.5kg/m2 ≤ body mass index (BMI) ≤ 35kg / m2, male weight ≥ 50kg, female weight ≥ 45kg.
3. Women of childbearing age need to be able to ensure effective contraception (medically approved contraceptive measures, such as intrauterine device, contraceptive pill or condom) during the trial and within 3 months after the end of the trial.
4. According to the diagnostic criteria of diagnostic and Statistical Manual of mental disorders (5th Edition) (dsm-5), it was diagnosed as severe depressive disorder, marked as moderate or severe, and without psychotic characteristics.
5. The total score of Montgomery Asperger Depression Scale (MADRS) in screening period and baseline was ≥ 22, and the CGI-S score was ≥ 4.
6. Compared with the screening period, the change in the total MADRS score at baseline did not exceed 25% of the screening period.
7. The patients fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the written informed consent, and are willing to complete the whole trial process according to the trial requirements.

Exclusion Criteria:

1. It meets dsm-5 diagnostic criteria for other mental disorders.
2. A depressive episode secondary to physical or other mental illness.
3. The researchers determined that there was a high risk of suicide: there were serious suicides and self injuries within 1 month before or during the screening; Or those who answered "yes" to item 5 of "suicidal ideation" in the screening Columbia suicide severity rating scale (c-ssrs).
4. The depressive episode is ineffective after sufficient treatment with one or more antidepressants (at least 6 weeks according to the dosage in the manual).
5. Those who had received electroconvulsive therapy (ECT) within 1 month before screening.
6. Patients who have received other stem cell therapy.
7. Have a history of infection within 1 month before screening and need hospitalization and / or antibiotic treatment; Or currently using systemic sex hormones (glucocorticoids), immunosuppressants or cytotoxic therapy.
8. Screening the patients who had been diagnosed with hyperthyroidism or hypothyroidism within the previous year and are still taking drugs; Or have a history of thyroid disease and thyroid stimulating hormone (TSH) is higher than 1.2 times the upper limit of normal value or lower than 0.8 times the lower limit of normal value;
9. Patients with a history of epilepsy (excluding children's history of fever and convulsion).
10. Persons with severe alcohol or drug dependence within 1 year before screening (excluding caffeine or nicotine); Or daily alcohol intake of or above 5 units (1 units =360mL wine or 45mL Baijiu or 120mL wine).
11. Accompanied by severe or unstable cardiovascular, respiratory, liver, kidney, blood, endocrine and central nervous system diseases.
12. Laboratory examination was abnormal, and the researcher determined that it was of important clinical significance, such as: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeded 2.5 times the upper limit of normal; Total bilirubin (TBIL) exceeds 1.5 times of the upper limit of normal value; Creatinine (CR) exceeded 1.2 times the upper limit of normal.
13. QTc interval of ECG in screening stage > 450 ms (male) or 470 MS (female); Or have a family history of long QT interval syndrome, or have cardiac insufficiency, severe arrhythmia or ischemic heart disease and need drug treatment, have congenital heart disease, severe organic heart disease or have a history of this disease.
14. HIV antibody, HBsAg, HCV antibody or syphilis serological test results are positive.
15. Participated in clinical trials of other drugs within 30 days before screening.
16. Pregnant or lactating women.
17. Patients with contraindications or allergies treated in this study.
18. The researcher considered that it was not suitable to participate in this experiment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The total score of Montgomery Asperger Depression Scale (MADRS) decreased from baseline after 8 weeks of treatment | 8 weeks

SECONDARY OUTCOMES:
Effective rate of treatment (effective: the total score of MADRS decreased by ≥ 50% compared with baseline) | 8 weeks
Remission rate of treatment (remission: MADRS total score ≤ 11 points) | 8 weeks

IPD SHARING:
Plan to Share IPD: No